CLINICAL TRIAL: NCT03793686
Title: A Phase 1 Double Blind, Randomized Clinical Study to Evaluate the Safety of Human Milk Oligosaccharides Following Antibiotic Therapy in Subjects With C. Difficile-associated Diarrhea
Brief Title: A Study of Safety of PBCLN-003 Following Antibiotic Therapy in Subjects With C.Difficile-associated Diarrhea
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18-CT-001
Record Dates: First submitted 2018-12-27; First posted 2019-01-04 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Clostridium Difficile Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PBCLN-003, daily in 3 divided oral doses for 7 days, 2 ascending dose cohorts
  Interventions: Drug: PBCLN-003
- Placebo (Placebo Comparator): Placebo, daily in 3 divided oral doses for 7 days, 2 ascending dose cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBCLN-003 — Investigational drug
  Arms: Experimental
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This Phase I double blind, randomized clinical study to evaluate the safety of human milk oligosaccharides (HMO) is designed to assess the safety and dosage ranging of PBCLN-003 in adults with Clostridium difficile-associated diarrhea (CDAD). Within 3 dose cohort, subjects will be randomized in a 3:1 ratio to receive PBCLN-003 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment episode of CDAD diagnosed based on > 3 loose stools per day and detection of CD toxin by nucleic acid amplification tests (NAAT), EIA or GDH
* Mild to moderate CDAD during enrollment episode (per Society of Hospital Epidemiologists of America (SHEA)/lnfectious Disease Society of America(ISDA) criteria)
* Current therapy with standard of care antibiotics for recurrent CDAD(vancomycin, metronidazole, fidaxomicin)
* BMI > 18.5 and < 40
* Age 18 years or older
* Agreement to adhere to the study protocol
* Informed consent is obtained
* Women who are capable of bearing children must have a negative pregnancy test at the time of screening
* Female subjects of childbearing potential must use birth control (defined as oral or injectable contraceptives, intrauterine devices, surgical sterilization or a combination of a condom and spermicide) during the study period and for up to 8 weeks after the first drug of study.

Exclusion Criteria:

* Severe CDAD during enrollment episode (per SHEA/ISDA criteria) characterized as follows:

  * History of five (5) or more recurrences of CDAD within the past 12 months prior to potential study enrollment
  * History of fecal microbiome transplant or other microbiome directed experimental intervention for CDAD
  * History (ever) of CD complicating inflammatory bowel disease (Crohn's disease, ulcerative colitis), or history of bowel resection surgery (other than uncomplicated appendectomy) or history of other infectious diarrhea or diarrhea of unknown etiology since the initial episode of CDAD
* Clinically immunocompromised due to any primary immune or autoimmune deficiency, as a result of chronic disease, cancer or medication used to treat these diseases
* Initiating a new diet or weight loss amounting to 10% within two weeks prior to date of study entry
* Enrolled in another clinical study for the therapy of CDAD or affecting nutritional management during the study period
* Enrolled or has been enrolled in another experimental (IND) study within two weeks prior to date of study entry
* Is pregnant or lactating
* History of swallowing difficulties, including dysphagia or odynophagia for liquids or solids
* Use of any Probiotics (any formulation) within the two weeks prior to date of study entry
* New, or a change in the consumption of the following prescription medications or over-the-counter (OTC) medications within two weeks prior to date of study entry:

  * Proton pump inhibitors (for example: Prilosec®, Nexium®)
  * Histamine-2 receptor antagonists (for example: Zantac®, Pepcid®)
* Consumption of the following prescription medications during the current enrollment episode: • Bezlotuxamab/Zinplava®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Characterization of Adverse Events in a dose escalation study of PBCLN-003 | Up to 8 Weeks
  Comparison of adverse event reporting and grading results between groups using physical exams, safety related blood tests, and urinalysis, adverse event reports, and subject complaint logs.

CONTACTS AND LOCATIONS:
Overall Officials: David J Rechtman, MD, Study Director — Vice President, Medical Affairs, Prolacta Bioscience
Locations (1):
- Infectious Disease Specialist, Idaho Falls, Idaho, United States

IPD SHARING:
Plan to Share IPD: No